CLINICAL TRIAL: NCT04383041
Title: Digital Collected Patient Reported Outcomes in a Diabetes Cohort
Brief Title: Study to Learn More About Outcomes Reported by Patients Suffering From Type 2 Diabetes Using a Digital Data Collection Tool
Acronym: DePRO
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21318
Record Dates: First submitted 2020-04-23; First posted 2020-05-11 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Type 2 Diabetes: Patients with Metformin containing prescription drugs will be eligible for participation and consecutively invited to study participation in their pharmacy.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Completing questionnaires via ePRO app from their own mobile devices

SUMMARY:
In this study researchers want to gain more information on patients who are treated with Metformin for their Type 2 Diabetes. Adult female and male patients with a prescription of a Metformin containing drug will be invited to the study in a public pharmacy after the decision for treatment with Metformin has been made by the treating physician. The pharmacist will provide interested participants access to a special phone App and participants are asked to complete via this phone App a questionnaire on their health situation with special focus on their Type 2 Diabetes. This includes questions on complications and self-care activities in relation to their diabetes, questions on quality of life and health history. There will be no extra visit to the treating doctor or a pharmacy. The study is aiming to have the questionnaire completed by 300 participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult female or male patient
* Valid prescription for a Metformin containing drug approved in Germany
* Decision to initiate treatment with Metformin was made by the treating physician as part of the routine treatment practice
* Signed informed consent

Exclusion Criteria:

- Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female and male patients with a valid prescription of a Metformin containing drug will be consecutively invited to the study in a public pharmacy after the decision for treatment with Metformin has been made by the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Summary of Diabetes Self-Care Activities for Diabetes and Kidney Disease (SDSCA) Score | Baseline
  The SDSCA measure is a brief self-report questionnaire of diabetes self-management. It assesses the number of days per week in which respondents engage in diabetes health-related behaviors in the areas of general diet, diabetes-specific diet, physical activity, blood-glucose testing, foot care, and smoking. Minimum score 0. Maximum score 77. Higher scores indicate better self care.

SECONDARY OUTCOMES:
Association between SDSCA score and demographic/ disease characteristics | Baseline
  Association of Summary of Diabetes Self-Care Activities for Diabetes and Kidney Disease (SDSCA) with demographic and disease characteristics
Acceptance of participation | Baseline
Adherence to documentation | Baseline
Health related Quality of Life-EuroQol five dimensions Questionnaire (EQ-5D) | Baseline
  Descriptive system of health-related quality of life states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression).
DTSQ Participation rate | Baseline
  Diabetes Treatment Satisfaction Questionnaire (DTSQ) Number of invited, participating and non-participating patients (reasons for non-acceptance of study participation)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many locations, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Mueller C, Schauerte I, Martin S, Irrgang V. Evaluation of Self-care Activities and Quality of Life in Patients With Type 2 Diabetes Treated With Metformin Using the 2D Matrix Code of Outer Drug Packages as Patient Identifier: the DePRO Proof-of-Concept Observational Study. JMIR Diabetes. 2022 May 24;7(2):e31832. doi: 10.2196/31832. PMID 35608887
- [Derived] Mueller C, Schauerte I, Martin S. Evaluation of Self-Care Activities and Quality of Life in Patients With Type 2 Diabetes Mellitus Treated With Metformin Using the 2D Matrix Code of Outer Drug Packages as Patient Identifier: Protocol for the DePRO Proof-of-Concept Observational Study. JMIR Res Protoc. 2021 Jan 11;10(1):e21727. doi: 10.2196/21727. PMID 33427685
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/